CLINICAL TRIAL: NCT03140033
Title: Sublingual Misoprostol Versus Placebo to Reduce Blood Loss During Elective Cesarean Delivery : A Randomized Controlled Study
Brief Title: Sublingual Misoprostol to Reduce Blood Loss During Elective Cesarean Delivery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Fathy, Resident of obstetrics and gynecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MFathy
Record Dates: First submitted 2017-04-24; First posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Hemorrhage Postpartum
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Ranitidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol oral tablets (Active Comparator): 79 women will recieve 400 micrograms of misoprostol ( misotac) sublingually and 20 IU of oxytocin at cord clamping
  Interventions: Drug: Misoprostol Oral Tablet
- Ranitidine oral tablets (Placebo Comparator): 79 women will recieve ranitidine oral tablets sublingually and 20 IU of oxytocin at cord clamping
  Interventions: Drug: Ranitidine Oral Tablet

INTERVENTIONS:
Drug: Misoprostol Oral Tablet — at cord clamping the patient will recieve 400 micrograms of misoprostol sublingually
  Other Names: Misotac
  Arms: Misoprostol oral tablets
Drug: Ranitidine Oral Tablet — at cord clamping the patient will recieve ranitidine sublingually
  Other Names: Ranitak
  Arms: Ranitidine oral tablets

SUMMARY:
Sublingual Misoprostol to Reduce Blood Loss During Elective Cesarean Delivery : A Randomized Controlled Trial

DETAILED DESCRIPTION:
This study aims to evaluate efficacy and safety of subligual misoprostol in reducing blood loss during cesarean section , a randomized double blinded prospective controlled trial conducted at Ain Shams maternity hospital . 158 women who fulfilled the inclusion criteria enrolled in this study .the patients randomized into two groups one of them will receive sublingual misoprostol 400 micrograms ( misotac )and the other will receive placebo( Ranitak ),all patients will subjected to history,physical examination,and investigations.preparation of patients (preload and antibiotics )according to hospital protocol.All C.S will be perfomed using spinal anaesthesia ,pfannenstiel incision of the skin ,open of abdomen in layers ,at cord clamping the patients will receive the medication sublingual and 20IU of oxytocin intravenous infusion simultaneous by the anesthesiologist,then close in anatomical layers.blood loss during C.S will be calculated following placental delivery to the end of surgery,and from the end of the operation to 6h after birth.the need for additional uterotonics agents,blood transfusion and adverse effects of the study drug will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies
* women booked for elective C.S
* full term pregnancies
* primi gravida or previous one delivery ( either by spontaneous vaginal delivery or C.S )

Exclusion Criteria:

* blood disorders
* multiple pregnancy
* placenta previa
* polyhydramnios
* marked maternal anemia
* contraindications to prostaglandin e.g history of asthma , allergy to misoprostol
* previous 2 or more C.S

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Blood loss during cesarean sections | through study completion, an average of 1 year
  Blood loss will be estimated by the anesthesiologist Using soaked towels and suction set after delivery of placenta

SECONDARY OUTCOMES:
Vaginal bleeding | through study completion, an average of 1 year
  Calculation of the amount of vaginal bleeding according to the number of soaked pads used after cesarea section for the 1st 6 hrs. Each soaked pad equal 50 cc
Change in blood pressure and pulse | through study completion, an average of 1 year
  Change in blood pressure and pulse before and after the cesarean section
Blood loss after 24 hr. | through study completion, an average of 1 year
  The allowable blood loss (ABL) =[ estimated blood volume ( EBV ) x (intial hematocrit (HI ) - final hematocrit (HF) ] / HI ( initial hematocrit)
Need for additional uterotonic agent | through study completion, an average of 1 year
  Need for additional uterotonic agent e.g oxytocin - methyl ergotamine
Need for blood transfusion | through study completion, an average of 1 year
  number of patients receiving blood transfusion
Need for surgical measures to stop bleeding | through study completion, an average of 1 year
  Need for surgical measures to stop bleeding e.g uterine artery ligation , B-lynch sutures or Hysterectomy
Side effects of misoprostol | through study completion, an average of 1 year
  Nausea, Vomiting or Diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Amr H YEHIA, MD,MRCOG, Study Director — Ain Shams University-Maternity Hospital
Locations (1):
- Ain shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes